CLINICAL TRIAL: NCT07139301
Title: Timing of Anticoagulation After Emergency Endovascular Therapy for Acute Ischemic Stroke With Atrial Fibrillation：a Randomised Controlled Trial
Brief Title: Timing of Anticoagulation After Emergency Endovascular Therapy for Acute Ischemic Stroke With Atrial Fibrillation
Acronym: TIMERS-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIMERS-1
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Stroke; Atrial Fibrillation
Keywords: Endovascular Therapy; Direct oral anticoagulation; Therapy initiation; Randomized Controlled Trial; Stroke
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early anticoagulation (Experimental): Early initiation of any direct oral anticoagulant (DOAC) within 96 hours (4 days) of the onset of acute ischemic stroke
  Interventions: Drug: Early anticoagulation
- Delayed anticoagulation (Active Comparator): Delayed initiation of any direct oral anticoagulant (DOAC) between 5-14 days of the onset of acute ischemic stroke
  Interventions: Drug: Delayed anticoagulation

INTERVENTIONS:
Drug: Early anticoagulation — Early initiation of direct oral anticoagulants will be started within four days after symptom onset.
  Arms: Early anticoagulation
Drug: Delayed anticoagulation — Delayed initiation of direct oral anticoagulants will be started between 5-14 days after symptom onset.
  Arms: Delayed anticoagulation

SUMMARY:
This study evaluates the safety and efficacy of early versus delayed initiation of direct oral anticoagulants (DOACs) in patients with acute ischemic stroke related to atrial fibrillation after emergency endovascular therapy (EVT).

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label, randomized controlled trial evaluating the safety and efficacy of different initiation timings of direct oral anticoagulants (DOACs) therapy in patients with acute ischemic stroke related to atrial fibrillation after emergency endovascular therapy (EVT).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or over.
2. Clinical diagnosis of large vessel occlusion acute ischemic stroke.
3. Emergency endovascular treatment was performed within 24 hours of stroke onset.
4. Atrial fibrillation (including paroxysmal, persistent or permanent atrial fibrillation), confirmed by at least one of the following:

   1. 12-lead ECG recording
   2. Inpatient ECG telemetry
   3. Prolonged ECG monitoring (e.g. Holter monitor)
   4. Previously established diagnosis of atrial fibrillation verified by medical records.
5. CT or MRI demonstrating one of the following findings:

   1. No hemorrhagic transformation;
   2. Hemorrhagic infarction type 1 (HI1), defined as small petechiae along the margins of the infarct (Heidelberg classification);
   3. Hemorrhagic infarction type 2 (HI2), defined as confluent petechiae within the infarcted area without space-occupying effect (Heidelberg classification).
6. Time from stroke onset to randomization was within 72 hours.
7. Written informed consent obtained from the patient or a legally authorized representative.

Exclusion Criteria:

1. Atrial fibrillation due to reversible causes (e.g. thyrotoxicosis, pericarditis, recent surgery, or myocardial infarct).
2. Contraindication to the use of direct oral anticoagulants (DOACs):

   1. Known allergy or intolerance to both factor Xa inhibitors and direct thrombin inhibitors;
   2. Definite indication for vitamin K antagonist (VKA) treatment (e.g. mechanical heart valve, valvular atrial fibrillation);
   3. Severe renal impairment (defined as creatinine exceeding 1.5 times of the upper limit of normal range) and significant hepatic dysfunction (defined as ALT or AST > twice the upper limit of normal range) ;
   4. Concomitant use of medications with significant interactions with DOACs, including azole antifungals, HIV protease inhibitors, or strong CYP3A4 inducers;
   5. Baseline platelet count < 100 x 109/L;
   6. History of coagulopathy or systemic hemorrhage.
3. Prior DOAC use within 48 hours of stroke onset, or recent treatment with vitamin K antagonist (VKA) leading to INR ≥1.7 at randomization.
4. Pregnant or breastfeeding women, or positive pregnancy test at admission.
5. History of major surgery or severe trauma within 1 month prior to stroke onset.
6. History of active bleeding within 1 month prior to stroke onset (e.g. gastrointestinal bleeding, urinary tract bleeding).
7. Dual antiplatelet therapy at baseline, or strong likelihood of requiring dual antiplatelet therapy during the trial.
8. Evidence of cerebral amyloid angiopathy.
9. CT or MRI evidence of non-stroke pathology likely to account for the presenting clinical symptoms (e.g. mass lesion, encephalitis).
10. Modified Rankin scale (mRS) score > 1 prior to stroke onset.
11. Inability to complete the 90-day follow-up.
12. Currently participating in another drug clinical trial.
13. Any other reason deemed by the investigator to make the patient unsuitable for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of recurrent ischemic stroke, symptomatic intracranial hemorrhage, and all-cause death | 90 days

SECONDARY OUTCOMES:
Incidence of recurrent ischemic stroke | 90 days
Incidence of venous thromboembolism | 90 days
Incidence of systemic embolism | 90 days
Incidence of myocardial infarction | 90 days
Proportion of Patients Achieving mRS 0-1 at 90 Days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Proportion of Patients Achieving mRS 0-2 at 90 Days | 90 days
  The modified Rankin scale (range, 0 [no symptoms] to 6 [death])
Length of hospital stay for stroke-related care | 90 days
Quality of life at 90 days assessed by EuroQol 5 Dimensions 5 level questionnaire [EQ-5D-5L] | 90 days
  The EQ-5D-5L includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicating worse quality of life.
Incidence of vascular death | 90 days
All-cause mortality | 90 days
Incidence of symptomatic intracranial haemorrhage (sICH) | 90 days
Incidence of major extracranial bleeding | 90 days

CONTACTS AND LOCATIONS:
Locations (40):
- China (40):
  - Ma'anshan People's Hospital, Ma’anshan, Anhui
  - Aviation General Hospital, Beijing, Beijing Municipality
  - Beijing Shijingshan Hospital, Beijing, Beijing Municipality
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - Heyuan People's Hospital, Heyuan, Guangdong
  - Qinzhou First People's Hospital, Qinzhou, Guangxi
  - Baoding Sixth Hospital, Baoding, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Hongda Hospital of Jiamusi University, Jiamusi, Heilongjiang
  - Fangcheng County People's Hospital, Nanyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Lushan County People's Hospital, Pingdingshan, Henan
  - Xinyang Central Hospital, Xinyang, Henan
  - Queshan County People's Hospital, Zhumadian, Henan
  - Tianyou Hospital, Wuhan University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Yingkou Central Hospital, Yingkou, Liaoning
  - Ordos Central Hospital, Ordos, Neimenggu
  - Feicheng Hospital Of Shandong Yiyang Health Group, Feicheng, Shandong
  - Jinan Zhangqiu District People's Hospital, Jinan, Shandong
  - Laizhou City People's Hospital, Laizhou, Shandong
  - Liaocheng Neurological Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Linshu County People's Hospital, Xiazhuang, Shandong
  - Yantai Yeda Hospital, Yantai, Shandong
  - Guoyao Northern Hospital (Baotou), Baotou, Shanxi
  - ShanXi Cardiovascular Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The People's Hospital of Yueqing, Yueqing, Zhejiang
  - Xuanwu Hospital, Beijing, Beijing 100053, Beijing
  - Guoluo Prefecture People's Hospital, Guoluo
  - Huanghua Municipal People's Hospital, Huanghua
  - First Affiliated Hospital of Henan Polytechnic University, Jiaozuo
  - Qilu Hospital of Shandong University, Jinan
  - Ningjin County People's Hospital, Ningjin
  - Ren Shou County People's Hospital, Renshou
  - Daliuta Experimental District People's Hospital of Shenmu City, Shenmu
  - Xiuyan Central Hospital, Xiuyan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou

IPD SHARING:
Plan to Share IPD: No
The study is proceeding.